CLINICAL TRIAL: NCT00957125
Title: PROMIX - Preoperative Treatment of Breast Cancer With a Combination of Epirubicin, Docetaxel and Bevacizumab. A Translational Trial on Molecular Markers and Functional Imaging to Predict Response Early. A Phase 2 Study.
Brief Title: A Translational Trial on Molecular Markers and Functional Imaging to Predict Response of Preoperative Treatment of Breast Cancer Early
Acronym: PROMIX
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Thomas Hatschek (Other)
Responsible Party: Sponsor-Investigator, Thomas Hatschek, MD, PhD, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROMIX; 2007-005858-23 (EudraCT Number)
Record Dates: First submitted 2009-08-10; First posted 2009-08-12 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
Keywords: Localized primary breast cancer; Inflammatory breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Epirubicin; Docetaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Epirubicin Docetaxel Bevacizumab (Experimental): Epirubicin and docetaxel i.v. infusion q 3 weeks for 2 cycles.
  * If complete response this treatment continues for 4 cycles, totally 6 cycles.
  * If partial response or stable disease, epirubicin and docetaxel and bevacizumab i.v. infusion q 3 weeks for 4 cycles.
  * If progressive disease after the first 2 cycles individualized treatment.
  Interventions: Drug: Epirubicin; Drug: Docetaxel; Drug: Bevacizumab

INTERVENTIONS:
Drug: Epirubicin — 75 mg/m2 i.v. infusion, 30 min, cycle day 1, cycles 1-6.
Drug: Docetaxel — 75 mg/m2 i.v. infusion, 60 min, cycles day 1, cycle 1-6.
  Other Names: Taxotere
Drug: Bevacizumab — 15 mg/kg, i.v. infusion, 90 min, cycle day 1, cycles 3-6 if PR or SD after cycle 2.
  Other Names: Avastin

SUMMARY:
Patients with localized primary breast cancer including inflammatory breast cancer suitable for primary medical treatment and/or regional lymph node metastases receive six cycles of chemotherapy with epirubicin and docetaxel. Treatment evaluations are performed after the second, fourth and sixth cycle. In case of SD/PR after the second course, bevacizumab is added to the combination for the remaining four courses.

Besides standard response evaluation clinically and by mammography and ultrasound, several functional imaging techniques including MR, CT-PET and contrast-enhanced ultrasound are investigated. Fresh tumor tissue samples from the primary tumor are collected before start, after two courses and in connection with surgery. The aim of the trial is to detect biological factors and functional imaging techniques with the ability to predict response at an early stage of treatment.

DETAILED DESCRIPTION:
Primary endpoints: Objective response (OR) characterized by conventional radiological and functional imaging procedures and biological tumour markers at an early point of treatment with epirubicin + docetaxel and effects of addition of bevacizumab as reflected by these procedures. Early functional and biological changes signalling pathological complete response (pCR). Secondary endpoints: Secondary endpoints: Morphological and biological changes of tumours exposed for cytotoxic and targeted treatment. Disease-free survival. Safety.

Evaluations:

Before start of treatment:

Tumour staging: Bone scan, chest X-ray and liver ultrasound or CT scan of chest and abdomen within four weeks before start of treatment. Physical examination, conventional radiology (ultrasound and mammography including pre-treatment localization with carbon suspension) and functional imaging procedure (MRI or PET-CT or Contrast-Enhanced Ultrasound (CEUS) or Scintigraphy with 99m-Tc-HMPAO (Ceretec)) within two weeks before start of treatment.

Blood samples (SNP, metabolomics, M-30 assay, TK/XPA-210 assay, angiogenesis markers, TIMP-1, tissue factor) and tumour biopsies (transcriptomics, proteomics, IHC-stroma, AMOT) are collected within two weeks before start of treatment.

During treatment:

Physical examination before start of each treatment. Imaging procedures: Mammography, ultrasound (compulsory) one week (5-9 days) after cycles 2, 4 and 6. MRI, PET-CT, Contrast-Enhanced Ultrasound (CEUS) applied according to availability at the participating sites, one week (5-9 days) after cycles 2 and 4.

Tumour markers: Blood samples (proteomics, metabolomics, M-30 assay, TK/XPA-210 assay, angiogenesis markers, TIMP-1, tissue factor) are collected 48 hours after cycles 1 thru 4. Tumour tissue (transcriptomics, proteomics, IHC-stroma, AMOT) is taken charge of by biopsy one week (5-9 days) after cycle 2 and from the tumour specimen in connection with surgery.

Totally, 150-200 patients with measurable/evaluable primary breast cancer are planned for inclusion within a period of two years time. For each imaging method, approximately 40-50 patients will be included. The study is designed to find early predictors of response by testing a set-up of several different molecular and imaging tools. In addition, for each method changes of patterns occurring during treatment will be compared to baseline findings and, in the case of functional imaging, standard imaging procedures.

All patients will be followed for five years after operation with regard to outcome and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Female patients with breast cancer confirmed by histology.
* Tumour and blood samples according to APPENDIX I available.
* Age 18 years or older. Elderly patients in condition adequate for chemotherapy.
* Localized primary breast cancer including inflammatory breast cancer suitable for primary medical treatment and/or regional lymph node metastases including ipsilateral supraclavicular nodes with breast cancer diagnosis confirmed by histological examination with or without breast tumour lesions.
* Adequate bone marrow, renal, hepatic and cardiac functions and no other uncontrolled medical or psychiatric disorders.
* ECOG performance status 0-1.
* Patients in child-bearing age with adequate contraception.

Exclusion Criteria:

* Distant metastases, including node metastases in the contralateral breast region and in the mediastina.
* Other malignancy for the last two years except for radically treated basal or squamous cell carcinoma of the skin or CIS of the cervix.
* HER2-amplification verified by FISH analysis.
* Pregnancy or lactation.
* Uncontrolled hypertension, heart, liver, kidney related or other medical or psychiatric disorders.
* Recent history of thromboembolism and ongoing medication with full-dose anticoagulants.
* Major surgery (including open biopsy), significant traumatic injury within 28 days prior to enrollment or anticipation of the need for major surgery during study treatment.
* Minor surgery, including insertion of an indwelling catheter, within 24 hours prior to the first bevacizumab infusion.
* History or evidence of inherited bleeding diathesis or coagulopathy with the risk of bleeding.
* Non-healing wound, active peptic ulcer or bone fracture.
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months of enrollment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2008-09; Primary Completion 2011-11 (Actual); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the sensitivity and of defined diagnostic and biological procedures to detect response/non-response to neoadjuvant treatment at an early point among patients with breast cancer. | 6 weeks

SECONDARY OUTCOMES:
Identification of tumour characteristics and treatment-related changes of tumour characteristics predictive of long-term prognosis. | 5 years
Comparison between the standard evaluation procedures mammography, conventional ultrasound and clinical examination and functional imaging techniques and biological procedures with emphasis on detection of response at an early point of treatment. | 6 weeks
Studies on the addition of bevacizumab with regard to further improvement of response in tumours with stable (SD) or partial response (PR) and the impact of treatment on angiogenesis and local features of the tumour environment. | 6 weeks
Acute toxicity | 6 weeks after last chemotherapy
Late toxicity | 5 years after last chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hatschek, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (6):
- Sweden (6):
  - Sahlgrenska University Hospital, Gothenburg
  - Lund University Hospital, Lund
  - Malmö General University Hospital, Malmo
  - Karolinska University Hospital, Dept of Oncology, Stockholm
  - County Hospital, Sundsvall
  - Uppsala University Hospital, Uppsala

REFERENCES:
- [Result] Saracco A, Szabo BK, Tanczos E, Bergh J, Hatschek T. Contrast-enhanced ultrasound (CEUS) in assessing early response among patients with invasive breast cancer undergoing neoadjuvant chemotherapy. Acta Radiol. 2017 Apr;58(4):394-402. doi: 10.1177/0284185116658322. Epub 2016 Jul 28. PMID 27461224
- [Derived] Tribukait B. Early prediction of pathologic response to neoadjuvant treatment of breast cancer: use of a cell-loss metric based on serum thymidine kinase 1 and tumour volume. BMC Cancer. 2020 May 18;20(1):440. doi: 10.1186/s12885-020-06925-y. PMID 32423477
- [Derived] Nakamura M, Zhang Y, Yang Y, Sonmez C, Zheng W, Huang G, Seki T, Iwamoto H, Ding B, Yin L, Foukakis T, Hatschek T, Li X, Hosaka K, Li J, Yu G, Wang X, Liu Y, Cao Y. Off-tumor targets compromise antiangiogenic drug sensitivity by inducing kidney erythropoietin production. Proc Natl Acad Sci U S A. 2017 Nov 7;114(45):E9635-E9644. doi: 10.1073/pnas.1703431114. Epub 2017 Oct 23. PMID 29078273
- See also: Swedish website of the study. Password required — http://www.kpeks.se/promix